CLINICAL TRIAL: NCT04827862
Title: RADVAX™ for Relapsed/Refractory Non-Hodgkin Lymphoma: A Phase II Trial of Pembrolizumab + Low Dose Radiotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 56419; 844686 (Other: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab and Radiation Therapy (Experimental): pembrolizumab plus low-dose (4 Gy x 5) involved-site radiotherapy
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — pembrolizumab plus low-dose (4 Gy x 5) involved-site radiotherapy

SUMMARY:
This study is an open-label Phase II trial of non-Hodgkin lymphoma patients receiving initial treatment with the immunomodulatory agent, pembrolizumab, plus low-dose (4 Gy x 5) involved-site radiotherapy. Eligible patients will have r/r disease with at least 2 sites of measurable disease (≥1.0 cm), and must be eligible for treatment with pembrolizumab. Biosamples (blood and, where available, tumor) will be collected as outlined below. Pembrolizumab will be continued after RT until disease progression, drug intolerance, or at the discretion of the treating medical oncologist.

ELIGIBILITY:
Inclusion Criteria:

- Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of relapsed/refractory non-Hodgkin lymphoma (defined below) will be enrolled in this study.

Male participants:

- A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.

Female participants:

- A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.

   - The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.

   - Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
   * Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
   * Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the start date of radiation.
   * Have adequate organ function as defined in the following table (Table 1). Specimens must be collected within 10 days prior to the start of study drug Pembrolizumab.

   Note: The patient can be considered eligible and started on RT prior to confirming adequate organ function is met provided they meet the rest of the eligibility criteria. Adequate organ function needs to be confirmed prior to starting the Pembrolizumab. If it is found that the patient does not have adequate organ function post starting RT and prior to administering Pembrolizumab they will be withdrawn from the study and considered as a screen failure.

   - Pathologically confirmed B-cell, T-cell, aggressive, or indolent non-Hodgkin lymphoma for whom pembrolizumab is clinically indicated per physician discretion as documented in a separate Medical Oncology note.

   - Relapsed/refractory disease treated with at least 2 lines of prior therapy.

   • Relapsed disease is defined as progression of disease after achieving a remission to the most recent therapy.

   • Refractory disease is defined as failure to achieve CR or PR.

   • At least 2 lines of prior therapy are required, but, at physician and patient discretion with shared decision-making, not all FDA-approved treatments need be exhausted prior to enrollment.
   * For DLBCL and PMBCL:

     * Have relapsed after auto-SCT or have failed to achieve a CR or PR within 60 days of auto-SCT. Patients may have received intervening therapy after auto-SCT for relapsed or refractory disease, in which case they must have relapsed after or be refractory to their last treatment.
     * For patients who are ineligible for auto-SCT, have received at least ≥ 2 lines of prior therapy and have failed to respond to or relapsed after their last line of treatment. For patients who received consolidative local radiotherapy after systemic therapy, local radiotherapy will not be considered as a separate line of treatment.
   * Prior chimeric antigen receptor T-cell (CART) therapy is allowed but not required.

     • If the patient has received CART therapy, complete resolution of any active cytokine release syndrome is required 13. ≥2 sites of measurable disease (≥1.0 cm), at least one outside of intended RT fields.

     14. Ability to provide written informed consent.

   Exclusion Criteria:
   * A WOCBP who has a positive urine pregnancy test within 72 hours prior to the first fraction of radiation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.

   A patient may be considered eligible pending negative pregnancy test within 72 hours prior to the first fraction of radiation.
   * Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137).
   * Has received prior systemic anti-cancer therapy including investigational agents within 2 weeks prior to the first fraction of radiation.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

   Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.

   - Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.

   - Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.

   - Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

   - Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.

   - Has a known additional malignancy that is progressing or has required active treatment within the past 1 year. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, breast cancer, prostate cancer, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.

   - Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.

   - Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

   - Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.

   - Has an active infection requiring systemic therapy.

   - Has a known history of active TB (Bacillus Tuberculosis).

   - Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

   - Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

   - Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

   - Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.

   - Has undergone allogeneic bone marrow transplantation within 5 years.
   * History of graft-versus-host-disease.
   * Has a known history of Human Immunodeficiency Virus (HIV).
   * Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
CR rate | 12 weeks

SECONDARY OUTCOMES:
Time to best response | 20 weeks
Duration of best response | 5 years
Progression-free survival (PFS) | 5 years
Overall survival | 5 years
Duration of immunotherapy use for the pembrolizumab + RT induction CR cohort | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael LaRiviere, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abamson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT04827862/Prot_SAP_000.pdf